CLINICAL TRIAL: NCT02145858
Title: Prevention of Retained-Blood Outcomes With Active Clearance Technology. ACT Registry
Brief Title: Prevention of Retained-Blood Outcomes With Active Clearance Technology
Status: Completed | Type: Observational
Sponsor: ClearFlow, Inc. (Industry)
Collaborators: Vanderbilt University Medical Center (Other); Catholic Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CL2014001
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Hemorrhage; Atrial Fibrillation, Postoperative
Keywords: atrial fibrillation, pericardial effusion, pleural effusion
MeSH Terms: conditions — Hemorrhage; Atrial Fibrillation; Pericardial Effusion; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Blood drainage post cardiac surgery using PleuraFlow System

SUMMARY:
Postoperative bleeding is a common consequence after heart surgery which can significantly impact outcomes and costs . When bleeding occurs, reliable postoperative blood evacuation of the pleural, mediastinal and pericardial spaces with chest tubes is imperative to facilitate pulmonary reexpansion and mediastinal decompression as the patient recovers. When postoperative blood evacuation is inadequate, complications from retained blood can result. Clinically, retained blood may be recognized acutely or sub acutely. The acute clinical presentation is usually blood and fresh thrombus around the heart or lungs presenting as tamponade or hemothorax. The subacute clinical presentation is bloody pleural or pericardial effusions. These effusions are often driven by the breakdown of remaining thrombus. Once retained blood occurs, subsequent procedures may be needed to remedy it. Interventions to remove postoperative pericardial and/or pleural fluid or blood and reoperations due to bleeding are captured under a composite termed Retained Blood Syndrome, or RBS. The need for treatment and interventions for these conditions represents an impediment to patient recovery and involves both resource and economic consumption for a heart program and the healthcare system at large.

A recent review of the literature indicates that additional procedures for RBS are demonstrated in approximately 15% to 20% of patients after heart surgery. In a prospectively collected US Nationwide Inpatient Sample (NIS) data from 2010, RBS could be demonstrated in 17% of patients. In this analysis, mortality was doubled from 4% to 8%, length of stay was increased by 5 days, and average costs were 55% higher. Patients with RBS, therefore, represent an increased at-risk population for complications and costs.

Postoperative obstruction of conventional chest tubes with blood and other fibrinous material in the setting of postoperative bleeding contributes to RBS. In a study of postoperative cardiac surgery patients at the Cleveland Clinic, 36% of patients were found to have evidence of chest tube obstruction. Active Clearance with PleuraFlow has been shown to prevent chest tube clogging, and reduce RBS.

The purpose of this registry is to evaluate the effectiveness of the PleuraFlow System, a commercial Class II (US), Class IIb (Canada, Europe, and Australia), in the management of blood evacuation after cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective multicenter observational registry with a retrospective control. The registry has two tracks. One track--ALL-ACT-- is for sites enrolling a consecutive cohort of all cardiac surgery patients (Track A). The second track--VAD-ACT-- is for sites enrolling patients post ventricular assist device (VAD) surgery (Track B). There are two conditions for participation in this registry:

First, sites are required to provide anonymized matched historical data elements from a cohort of cardiac surgery patients done over the preceding 12 to 24-month period (Phase 0). These retrospective data elements will be used as baseline information for the purpose of comparative analyses (control group) with the prospective data sets collected during the prospective enrollment phase (treatment group).

Second, sites are required to participate in a roll-in phase (Phase 1). The purposes of the roll-in phase are to allow the users at participating sites to familiarize themselves with the use of the product with Active Clearance Technology; to implement clinical use protocols provided by ClearFlow, Inc. to all commercial users as part of product training, and; to demonstrate consistency and compliance with the clinical use protocols.

Phase 0 and phase 1 can be executed in parallel. Participating sites may start prospective enrollment (Phase 2) after completion of phase 0 and 1.

Investigators shall report PleuraFlow-related serious injuries to Sponsor as soon as becoming aware of the injury and no later than 48 hours.

Investigators shall report deaths to both the Sponsor and Regulatory authorities in compliance with their applicable State, Country and conditions imposed by the reviewing Ethical Committee. The three main guidance documents for reporting recall and vigilance procedure of medical devices are, 21 CFR, Part 806, MEDDEV 2.12/1 rev8 Guidelines on a Medical Devices Vigilance System, and Health Canada Medical Device Regulations SOR/98-282.

Vanderbilt University will create a REDCap database specific to this study and administer it. The Vanderbilt database study administrator will control database access, oversee data entry and data transfer from each participating site. Database manager will monitor the REDCap database and ensure data completeness and security. The database manager will maintain contact will the data entry personnel from each site and ensure whether data capture is occurring and determine the number of patients expected to be enrolled in the Registry at the end of the study period. Sponsor will not have access to REDCap once the study is complete. The REDCap database is secure and HIPAA compliant.

Descriptive statistics for categorical variables will be reported as percentages, and continuous variables will be reported as mean ± standard deviation (SD). Categorical variables will be compared using the chi-square test. Continuous variables will be compared using a Student's t-test as appropriate.

Database study administrator will coordinate the generation of data reports and statistical outputs. Sponsor will not have access to REDCap once the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects 18 years or older who received a PleuraFlow System following heart surgery.
* Patient undergoing cardiac surgery via sternotomy.

Exclusion Criteria:

* Any condition deemed inappropriate for inclusion by the investigators.
* Infants, children and adolescents under the age of 18.
* Robotic surgery.
* Any access via thoracotomy.
* Intolerance to implantable silicone materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older who received a PleuraFlow System following heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Retained Blood Syndrome (RBS) | surgery to post-operative 30 days
  The incidence of RBS as defined by a composite endpoint of specific interventions and diagnoses. Any patient that has a record of any of the following interventions or diagnoses post-operatively including post-discharge, will be considered to have RBS.
  * Interventions
    * Reoperation for bleeding, tamponade or washout of retained blood
    * Pericardial window
    * Chest tube placement/replacement
    * Pericardiocentesis
    * Placement of pericardial drain
    * Thoracotomy
    * Thoracoscopy
    * Thoracentesis
  * Diagnoses
    * Pleural effusion
    * Pericardial effusion
    * Hemothorax
    * Pneumothorax
    * Pericardial tamponade

CONTACTS AND LOCATIONS:
Overall Officials: Simon Maltais, MD, Study Director — Mayo Clinic, Rochester, MN
Locations (2):
- United States (2):
  - Catholic Medical Center, Manchester, New Hampshire
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Boyle EM Jr, Gillinov AM, Cohn WE, Ley SJ, Fischlein T, Perrault LP. Retained Blood Syndrome After Cardiac Surgery: A New Look at an Old Problem. Innovations (Phila). 2015 Sep-Oct;10(5):296-303. doi: 10.1097/IMI.0000000000000200. PMID 26575376
- [Background] Light RW. Pleural effusions following cardiac injury and coronary artery bypass graft surgery. Semin Respir Crit Care Med. 2001 Dec;22(6):657-64. doi: 10.1055/s-2001-18802. PMID 16088710
- [Background] Light RW. Pleural effusions after coronary artery bypass graft surgery. Curr Opin Pulm Med. 2002 Jul;8(4):308-11. doi: 10.1097/00063198-200207000-00011. PMID 12055394
- [Background] Light RW, Rogers JT, Cheng D, Rodriguez RM. Large pleural effusions occurring after coronary artery bypass grafting. Cardiovascular Surgery Associates, PC. Ann Intern Med. 1999 Jun 1;130(11):891-6. doi: 10.7326/0003-4819-130-11-199906010-00004. PMID 10375337
- [Background] Light RW, Rogers JT, Moyers JP, Lee YC, Rodriguez RM, Alford WC Jr, Ball SK, Burrus GR, Coltharp WH, Glassford DM Jr, Hoff SJ, Lea JW 4th, Nesbitt JC, Petracek MR, Starkey TD, Stoney WS, Tedder M. Prevalence and clinical course of pleural effusions at 30 days after coronary artery and cardiac surgery. Am J Respir Crit Care Med. 2002 Dec 15;166(12 Pt 1):1567-71. doi: 10.1164/rccm.200203-184OC. Epub 2002 Oct 11. PMID 12406850
- [Background] Ikaheimo MJ, Huikuri HV, Airaksinen KE, Korhonen UR, Linnaluoto MK, Tarkka MR, Takkunen JT. Pericardial effusion after cardiac surgery: incidence, relation to the type of surgery, antithrombotic therapy, and early coronary bypass graft patency. Am Heart J. 1988 Jul;116(1 Pt 1):97-102. doi: 10.1016/0002-8703(88)90255-4. PMID 3260740
- [Background] Shalli S, Boyle EM, Saeed D, Fukamachi K, Cohn WE, Gillinov AM. The active tube clearance system: a novel bedside chest-tube clearance device. Innovations (Phila). 2010 Jan;5(1):42-7. doi: 10.1097/IMI.0b013e3181cf7ce3. PMID 22437275
- [Background] Karimov JH, Gillinov AM, Schenck L, Cook M, Kosty Sweeney D, Boyle EM, Fukamachi K. Incidence of chest tube clogging after cardiac surgery: a single-centre prospective observational study. Eur J Cardiothorac Surg. 2013 Dec;44(6):1029-36. doi: 10.1093/ejcts/ezt140. Epub 2013 Mar 21. PMID 23520232
- [Background] Shiose A, Takaseya T, Fumoto H, Arakawa Y, Horai T, Boyle EM, Gillinov AM, Fukamachi K. Improved drainage with active chest tube clearance. Interact Cardiovasc Thorac Surg. 2010 May;10(5):685-8. doi: 10.1510/icvts.2009.229393. Epub 2010 Feb 23. PMID 20179137
- [Background] Arakawa Y, Shiose A, Takaseya T, Fumoto H, Kim HI, Boyle EM, Gillinov AM, Fukamachi K. Superior chest drainage with an active tube clearance system: evaluation of a downsized chest tube. Ann Thorac Surg. 2011 Feb;91(2):580-3. doi: 10.1016/j.athoracsur.2010.10.018. PMID 21256318
- [Background] Perrault LP, Pellerin M, Carrier M, Cartier R, Bouchard D, Demers P, Boyle EM. The PleuraFlow Active Chest Tube Clearance System: initial clinical experience in adult cardiac surgery. Innovations (Phila). 2012 Sep-Oct;7(5):354-8. doi: 10.1097/IMI.0b013e31827e2b4d. PMID 23274869
- [Background] Sirch J, Ledwon M, Puski T, Boyle EM, Pfeiffer S, Fischlein T. Active clearance of chest drainage catheters reduces retained blood. J Thorac Cardiovasc Surg. 2016 Mar;151(3):832-838.e2. doi: 10.1016/j.jtcvs.2015.10.015. Epub 2015 Oct 22. PMID 26611748
- [Derived] Baribeau Y, Westbrook B, Baribeau Y, Maltais S, Boyle EM, Perrault LP. Active clearance of chest tubes is associated with reduced postoperative complications and costs after cardiac surgery: a propensity matched analysis. J Cardiothorac Surg. 2019 Nov 8;14(1):192. doi: 10.1186/s13019-019-0999-3. PMID 31703606
- [Derived] Maltais S, Davis ME, Haglund NA, Perrault L, Kushwaha SS, Stulak JM, Boyle EM. Active Clearance of Chest Tubes Reduces Re-Exploration for Bleeding After Ventricular Assist Device Implantation. ASAIO J. 2016 Nov/Dec;62(6):704-709. doi: 10.1097/MAT.0000000000000437. PMID 27556153